CLINICAL TRIAL: NCT06728735
Title: Role of Next Generation Sequencing in the Etiological Diagnosis of Permanent Congenital Hypothyroidism with in Situ Thyroid: Preliminary Data in Patients Followed At the Regional Neonatal Screening Centre for Endrocrine-Metabolic Disease in Bologna
Brief Title: Role of Next Generation Sequencing in the Etiological Diagnosis of Permanent Congenital Hypothyroidism with in Situ Thyroid
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: IPOGEN2-20
Record Dates: First submitted 2024-12-03; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-10

CONDITIONS: Congenital Hypothyroidism
Keywords: Congenital Hypothyroidism
MeSH Terms: conditions — Congenital Hypothyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Retro-prospective, exploratory, single-centre observational study conducted at the Endrocrine-Metabolic Diseases Centre of the Pediatrics Unit, IRCCS Azienda Ospedaliero-Universitaria di Bologna, Italy.

The primary aim is to assess, by NGS sequencing of a panel of target genes, the frequency and type of variants with potential pathogenic significance in a patient population with congenital hypothyroidism and in situ thyroid, born between January 2003 and December 2023 identified through Neontal Screening at the Regional Centre for Neonatal Screening for Endrocrine-Metabolic Diseases, IRCCS Azienda Ospedaliero-Universitaria di Bologna, Italy.

DETAILED DESCRIPTION:
The primary aim of this study is to assess by NGS sequencing of a panel of target genes, the frequency and type of variants with potential pathogenic significance in a patient population with congenital hypothyroidism and in situ thyroid, born between January 2003 and December 2023 identified through Neontal Screening at the Regional Centre for Neonatal Screening for Endrocrine-Metabolic Diseases, IRCCS Azienda Ospedaliero-Universitaria di Bologna, Italy.

The secondary aims are to identify possible associations between genotype and phenotype; assess the risk of familial recurrence by searching for specific familial mutations; estimate the frequency of congenital hypothyroidisms with thyroid in situ out of the total number of congenital hypothyroidisms at the time of diagnostic confirmation; estimate the percentage frequency of transient and permanent congenital hypothyroidisms in patients with a thyroid in situ at diagnostic re-evaluation; identify possible prognostic factors for transient or permanent congenital hypothyroidism.

The retrospective phase of the study consists of the collection and analysis of clinical, hormonal and instrumental data of the cohort of patients enrolled by consulting their clinical records. More in detail, data on complete medical history, family history, physical examination with evaluation of major associated malformations, and thyroid ecography will be retrospectively collected.

Among this cohort, patients who have been diagnosed with permanent congenital hypothyroidism following diagnostic re-evaluation, according to clinical practice, will undergo molecular analysis by NGS sequencing of a panel of target genes for thyroid pathology.

ELIGIBILITY:
Inclusion Criteria:

* Patients born in Emilia-Romagna region, Italy, between January 2003 and December 2023;
* Patients screened at the Regional Neonatal Screening Centre for Endrocrine-Metabolic Diseases, IRCCS Azienda Ospedaliero-Universitaria of Bologna, Italy, and recalled for suspected congenital hypothyroidism;
* Confirmed diagnosis of congenital hypothyroidism and in situ thyroid;
* Hormonal and clinical follow-up of at least 36 months at Centre for Endrocrine-Metabolic Diseases, IRCCS Azienda Ospedaliero-Universitaria of Bologna, Italy;
* Obtaining informed consent from parents/legal guardians of paediatric patients.

Exclusion Criteria:

• Patients with hypothyroidism associated with chromosomal syndromes.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients born in Emilia-Romagna, Italy, between January 2003 and December 2023, recalled by the Regional Centre for Neonatal Screening for Endrocrine-Metabolic Diseases, IRCCS Azienda Ospedaliero-Universitaria di Bologna, Italy, for suspected congenital hypothyroidism and diagnosed with congenital hypothyroidism and in situ thyroid.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2021-03-17 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
NGS sequencing of a panel of target genes for thyroid pathology | At the time of diagnostic reevaluation, on average 1 year after diagnosis, if permanent congenital hypothyroidism is confirmed
  DUOX2, DUOXA2, FOXE1, GLIS3, IGSF1, IYD, NIKX2-1, NIKX2-5, PAX8, SLC16A2, SLC26A4, SLC5A5, TG, THRA, THRB, TPO, TSHB, and TSHR genes

SECONDARY OUTCOMES:
TSH value at screening test, and at diagnostic confirmation | at baseline
  microU/ml
ft4 values at diagnostic confirmation | at baseline
  pg/ml

CONTACTS AND LOCATIONS:
Overall Officials: Valeria Di Natale, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy